CLINICAL TRIAL: NCT03338829
Title: Incentive Models on Testing Adherence for Women With Diabetes During Pregnancy
Brief Title: Incentives and Glucose Adherence in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201603724
Record Dates: First submitted 2017-10-26; First posted 2017-11-09 (Actual); Results first posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Diabetes in Pregnancy
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): The control arm will receive compensation at time of enrollment for agreeing to participate.
- Positive Incentive (Experimental): The positive incentive arm will receive compensation per prescribed test, payable every month based on testing adherence.
  Interventions: Behavioral: Positive incentive
- Loss Aversion (Experimental): The loss aversion arm will have compensation deposited into a University of Iowa Women's Health account. The participant will then "lose" compensation depending on actual adherence to recommended testing
  Interventions: Behavioral: Loss aversion

INTERVENTIONS:
Behavioral: Positive incentive — Compensation is paid for each glucose test completed
  Arms: Positive Incentive
Behavioral: Loss aversion — Fixed compensation is offered to patients and they can earn a range of compensation at the completion of pregnancy depending on overall glucose testing adherence
  Arms: Loss Aversion

SUMMARY:
Diabetes in pregnancy carries significant pregnancy specific risks and requires frequent glucose monitoring to reduce these risks. This project compares the effect of two incentive schemes on adherence rates of glucose testing in pregnancy.

DETAILED DESCRIPTION:
Diabetes in pregnancy is associated with increased risks of maternal and fetal complications and can be challenging to manage due to increasing insulin requirements with advancing gestational age. Based on standard of care guidelines, patients with diabetes check their blood glucose at least 4 times per day. Optimal management requires frequent glucose self-monitoring and active management of abnormal blood sugars and medications by clinicians. Poorly controlled diabetes has both significant maternal and neonatal consequences: Improving test adherence could benefit both the pregnant woman and her fetus. In this study, we propose to test the effect of two incentive schemes on rates of glucose monitoring on pregnant women with diabetes requiring medication.

Pregnant women with diabetes requiring medication are invited to participate if they meet specific inclusion criteria (<29 weeks) and followed in our outpatient clinic. Participants are randomized into one of three groups:

1. control group - receive compensation at time of enrollment,
2. positive incentive group - receive compensation per test completed
3. loss aversion group - receive between a range of compensation depending on their overall level of adherence.

Primary outcome of the study is frequency of prescribed glucose testing in pregnancy

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with insulin dependent diabetes prior to 29 weeks gestation.

Exclusion Criteria:

* incarcerated, not English speaking

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women eligible
Enrollment: 130 (Actual)
Dates: Start 2016-05-05 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Andrews, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospital and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wernimont SA, Sheng JS, Tymkowicz A, Fleener DK, Summers KM, Syrop CH, Andrews JI. Adherence to self-glucose monitoring recommendations and perinatal outcomes in pregnancies complicated by diabetes mellitus. Am J Obstet Gynecol MFM. 2019 Aug;1(3):100031. doi: 10.1016/j.ajogmf.2019.100031. Epub 2019 Aug 5. PMID 33345801
- [Background] Homko CJ, Reece EA. Self-monitoring of blood glucose in gestational diabetes. J Matern Fetal Neonatal Med. 2002 Dec;12(6):389-95. doi: 10.1080/jmf.12.6.389.395. PMID 12683649
- [Background] de Veciana M, Major CA, Morgan MA, Asrat T, Toohey JS, Lien JM, Evans AT. Postprandial versus preprandial blood glucose monitoring in women with gestational diabetes mellitus requiring insulin therapy. N Engl J Med. 1995 Nov 9;333(19):1237-41. doi: 10.1056/NEJM199511093331901. PMID 7565999
- [Background] Halpern SD, French B, Small DS, Saulsgiver K, Harhay MO, Audrain-McGovern J, Loewenstein G, Brennan TA, Asch DA, Volpp KG. Randomized trial of four financial-incentive programs for smoking cessation. N Engl J Med. 2015 May 28;372(22):2108-17. doi: 10.1056/NEJMoa1414293. Epub 2015 May 13. PMID 25970009
- [Background] Sen AP, Sewell TB, Riley EB, Stearman B, Bellamy SL, Hu MF, Tao Y, Zhu J, Park JD, Loewenstein G, Asch DA, Volpp KG. Financial incentives for home-based health monitoring: a randomized controlled trial. J Gen Intern Med. 2014 May;29(5):770-7. doi: 10.1007/s11606-014-2778-0. Epub 2014 Feb 13. PMID 24522623
- [Background] Yee LM, McGuire JM, Taylor SM, Niznik CM, Simon MA. "I Was Tired of All the Sticking and Poking": Identifying Barriers to Diabetes Self-Care Among Low-Income Pregnant Women. J Health Care Poor Underserved. 2015 Aug;26(3):926-40. doi: 10.1353/hpu.2015.0073. PMID 26320923
- [Background] Higgins ST, Washio Y, Heil SH, Solomon LJ, Gaalema DE, Higgins TM, Bernstein IM. Financial incentives for smoking cessation among pregnant and newly postpartum women. Prev Med. 2012 Nov;55 Suppl(Suppl):S33-40. doi: 10.1016/j.ypmed.2011.12.016. Epub 2011 Dec 27. PMID 22227223
- [Background] Cosson E, Baz B, Gary F, Pharisien I, Nguyen MT, Sandre-Banon D, Jaber Y, Cussac-Pillegand C, Banu I, Carbillon L, Valensi P. Poor Reliability and Poor Adherence to Self-Monitoring of Blood Glucose Are Common in Women With Gestational Diabetes Mellitus and May Be Associated With Poor Pregnancy Outcomes. Diabetes Care. 2017 Sep;40(9):1181-1186. doi: 10.2337/dc17-0369. Epub 2017 Jul 19. PMID 28724718
- [Background] Tappin D, Bauld L, Purves D, Boyd K, Sinclair L, MacAskill S, McKell J, Friel B, McConnachie A, de Caestecker L, Tannahill C, Radley A, Coleman T; Cessation in Pregnancy Incentives Trial Team. Financial incentives for smoking cessation in pregnancy: randomised controlled trial. BMJ. 2015 Jan 27;350:h134. doi: 10.1136/bmj.h134. PMID 25627664
- [Derived] Wernimont SA, Fleener D, Summers KM, Deonovic B, Syrop CH, Andrews JI. The Effect of Financial Incentives on Adherence to Glucose Self-Monitoring during Pregnancy among Patients with Insulin-Requiring Diabetes: A Randomized Clinical Trial. Am J Perinatol. 2024 May;41(S 01):e259-e266. doi: 10.1055/a-1889-7765. Epub 2022 Jul 1. PMID 35777732

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: The control arm will receive $25.00 at time of enrollment for agreeing to participate.
- Positive Incentive: The positive incentive arm will receive $0.10 per prescribed test, payable every month based on testing adherence. For those with type 2 diabetes, the maximum daily payment will be $0.40. For those with type 1 diabetes , the maximum payment will be $0.70 per day.
  Positive incentive: Compensation is paid for each glucose test completed
- Loss Aversion: The loss aversion arm will have $100 deposited into a University of Iowa Women's Health account. The participant will then "lose" compensation depending on actual adherence to recommended testing.
  For 95% or more adherence, no money will be lost. For 85-94% adherence, $25 will be removed from account. For 70-84% adherence, $50 will be removed from account. For less than 69% adherence, $75 will be removed.
  Loss aversion: Fixed compensation is offered to patients and they can earn a range of compensation at the completion of pregnancy depending on overall glucose testing adherence
Period: Overall Study
Arm/Group | Control | Positive Incentive | Loss Aversion
Started | 42 | 43 | 45
Completed | 37 | 39 | 41
Not Completed | 5 | 4 | 4
Not completed — Lost to Follow-up | 4 | 2 | 4
Not completed — Pregnancy loss | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Positive Incentive | Control | Loss Aversion | Total
Number analyzed (Participants) | 39 | 37 | 41 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (0.79) | 31 (0.92) | 32 (0.93) | 31 (0.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 37 | 41 | 117
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Self-reported in electronic health record
  Participants
    Race/Ethnicity: White | 26 | 28 | 30 | 84
    Race/Ethnicity: Black | 7 | 4 | 7 | 18
    Race/Ethnicity: Hispanic/Latina | 3 | 4 | 3 | 10
    Race/Ethnicity: Asian | 1 | 0 | 1 | 2
    Race/Ethnicity: Multiracial | 2 | 1 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 37 | 41 | 117

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Glucose Monitoring
Description: Patients with type 1 diabetes were advised to monitor glucose seven times daily (fasting, 1hour post breakfast, pre- lunch, 1 hour post lunch, pre-dinner and 1 hour post dinner and nightly). Patients with type 2 and gestational diabetes were advised to have four glucose tests daily (fasting and 1hour post breakfast, lunch and dinner). Adherence to glucose testing was determined by the number of tests daily divided by the # of recommended tests daily and averaged over the course of the study as previously described
Time Frame: Pregnancy
Measure: Mean (Standard Error); unit: percentage of overall adherence
Arm/Group | Control | Positive Incentive | Loss Aversion
Number analyzed (Participants) | 37 | 39 | 41
percentage of overall adherence | 57.31 (5.12) | 58.48 (4.60) | 69.08 (3.75)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Control | Positive Incentive | Loss Aversion
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/39 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/39 | 0/41
Other Adverse Events (participants affected / at risk) | 0/37 | 0/39 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/29/NCT03338829/Prot_SAP_000.pdf